CLINICAL TRIAL: NCT01604746
Title: Open-label Phase 3b Study to Investigate the Safety of Ross River Virus (RRV) Vaccine From 6 to 12 Months After the Third Vaccination in Healthy Adults (Follow up to Precursor Study 880801)
Brief Title: Additional 6-Month Safety Follow-up After Completion of Precursor Study 880801
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 881201
Record Dates: First submitted 2012-05-19; First posted 2012-05-24 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Prophylaxis of Ross River Virus Infection
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Safety assessment (No Intervention): Vaccine safety will be assessed in the period between 6 and 12 months after the 3rd vaccination in precursor Study 880801 based on diaries distributed to all subjects for documentation of SAEs or AESI. Females who became pregnant after the 3rd vaccination in Study 880801 will be followed until end of pregnancy.
  Interventions: Biological: Ross River Virus (RRV) Vaccine

INTERVENTIONS:
Biological: Ross River Virus (RRV) Vaccine — Not applicable, no vaccine will be administered in this study. The RRV vaccine was administered in the precursor study.

SUMMARY:
The purpose of this study is to verify the long-term safety of a 2.5 µg, adjuvanted (aluminium hydroxide) dose of Ross River Virus (RRV) vaccine.

ELIGIBILITY:
Inclusion Criteria:

Subjects who participated in precursor Study 880801 and meet all of the following criteria:

* Subject received 3 RRV vaccinations in Study 880801
* Subject has completed Visit 6 in Study 880801
* Subject and, if applicable, subject´s parent(s)/legal guardian(s), understand the nature of the study and its procedures, agree to its provisions and provide written informed consent prior to study entry
* Subject provides written assent according to his/her age, if applicable

Exclusion Criteria:

* Subject has participated in another clinical study other than Study 880801 involving an investigational product (IP) or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1146 (Actual)
Dates: Start 2012-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Incidence of SAEs and AESI, such as arthritis, Guillain Barré Syndrome (GBS), encephalitis, convulsions, Bell´s palsy, neuritis, vasculitis, demyelinating disorders (ADEM and myelitis) and vaccination failure | 12 months after the third vaccination administered in precursor study 880801
  SAE = Serious adverse event, AESI = Adverse event of special interest

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Aichinger, MD, Study Director — Baxter Innovations GmbH
Locations (13):
- Australia (13):
  - Holdsworth House Medical Practice, Darlinghurst, New South Wales
  - St. Vincent´s Hospital, Darlinghurst, New South Wales
  - National Centre for Immunisation Research & Surveillance, The Children´s Hospital Westmead, Westmead, New South Wales
  - Wesley Research Institute Clinical Trials Centre, The Wesley Hospital, Auchenflower, Queensland
  - Cairns Base Hospital, Cairns, Queensland
  - QPID Clinical Trials Centre, Royal Children´s Hospital, Herston, Queensland
  - Dept of Microbiology & Infectious Diseases, Bedford Park, South Australia
  - CMAX, a Division of the Institute of Drug Technology (IDT) Australia, Ltd., North Adelaide, South Australia
  - Barwon Health - The Geelong Hospital, Dept Clinical & Biomedical Sciencesl, Geelong, Victoria
  - Centre for Clinical Studies, Heidelberg, Victoria
  - Emeritus Research, Malvern East, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia